CLINICAL TRIAL: NCT03532321
Title: Stress at Work and Infectious Risk in Patients and Caregivers
Acronym: STRIPPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Conservatory of Arts and Crafts (Cnam) of Paris (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI16020J
Record Dates: First submitted 2018-02-07; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-01

CONDITIONS: Occupational Exposure to Blood; Healthcare-associated Related Infections; Stress; Fatigue
Keywords: Stress; occupational risks; hospital organization; longitudinal
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers: Caregivers in the participating hospital departments : medical (doctors, midwives) and paramedical (nurses' aides, registered nurses, specialized nurses and head nurses) staff, working in hospital departments drawn at random among five volunteer hospital centers in Paris, and who will be present at the time of investigator's passage, at a date drawn at random during the inclusion phase.
  Interventions: Other: NA : non interventional study

INTERVENTIONS:
Other: NA : non interventional study — NA : non interventional study

SUMMARY:
In hospitals, the improvement of working conditions is often considered secondarily to patient satisfaction. Previous studies, showing statistically significant relationships, suggested the impact of hospital departments' organization (staff / patient ratio, bed distribution, caregiver's assignment), of the work environment, and the working conditions on the infectious risk at the hospital departments. In addition, organizational hospital constraints and the organization of care could equally have a major impact on the physical and psychological health of care workers (stress, fatigue, job satisfaction). To date, available data suggest that determinants of occupational stress and fatigue are multifactorial.

This research aims to develop an interdisciplinary approach to link two phenomena that are often studied independently while they are closely intertwined: working conditions and infectious risk in hospitals departments. Their main objective is to study the relationship between stress and caregiver fatigue at the work, organizational determinants and infectious risk for patients (healthcare-associated infections: HAIs) and for caregivers (blood exposure accidents: BEAs). The secondary objective is to analyze how the individual characteristics of the staff, the characteristics of their employment, and the overall organization in the hospital departments where they work interact to explain their physical and psychological state of health, on the one hand, and their behavior face to work (absenteeism, turnover and hand hygiene) on the other hand. The ultimate goal of this research is to be able to propose organizational strategies aimed at both reducing the probability of occurrence of healthcare-associated infections and preventing occupational risks for caregivers.

DETAILED DESCRIPTION:
STRIPPS is an etiologic, multi-center cohort study in the Ile-de-France region aiming to study better understands the complex relationship between the work organization, the stress ant and the caregiver fatigue and infectious risk in the hospital departments.

It will be conducted in 5 volunteer hospitals, with 7 to 8 hospital departments selected at random in each center and meeting eligibility inclusion criteria. The envisaged recruitment is approximately 20 staff per hospital department, enabling a total of about 150 staff to be included per center, totaling 750 surveyed caregivers.

The five voluntary centers will designate at least one local correspondent or referent among the hygiene team, the human resources (HR) department and the department of medical information system (DMI). The hygiene referent is the privileged correspondent. He will be part of the scientific committee and will help the investigators in the organization of the study within the hospital departments that will be drawn to participate. The HR and DMI referents are appointed to facilitate the collection of anonymous and aggregated data from the HR and PMSI databases planned for the study.

After obtaining regulatory authorizations, the eligible hospital departments of each hospital center will be drawn at random. Prior to the draw, hygiene referents of each hospital will prepare a list with all eligible hospital departments. Hospital departments will be selected using simple random sampling without replacement as follows in each list, the services will be numbered from 1 to n and 8 numbers between 1 and n will be chosen randomly using a computer. It will have a total of 5 lists (one list per hospital center) and 8 randomly selected numbers per list for a total of 40 randomly selected services. Similarly, visit days and survey start schedules will be drawn at random for the passage of an epidemiologist investigator recruited by the coordinating team. Two survey dates, between one Monday and one Friday of each week, and one survey start schedule, will be drawn at random for each work shift in every participating hospital department, during the entire inclusion period. Information meetings with the staff of the selected participating hospital departments and the communication by display will be organized by the investigators. A 15-day period will be left between the last information meeting held in the service and the closest date drawn for the start of the inclusion visits.

Based on a prospective data collection and using a qualitative-quantitative approach this study will provide some elements to better understand the complex relationship between the work organization, the stress and the caregiver fatigue, and infectious risk in the hospital departments (for patients and caregivers). This is an approach that relies on a conceptual model with several hypotheses to test. The conceptual diagram envisaged in our study has been based on the James Reason's model of accident causation. Indeed, it considers a multi-level interrelation of many factors ranging from organizational climate root causes to infectious risk. This equally includes contributory factors related to caregivers themselves, the care team, work environment as well as immediate causes related to care practices. Thus, for example, the infectious risk such as blood exposure accidents (for caregivers) or healthcare-associated infections (for patients) could be explained by several relationships between a wide range of factors: behavioral changes in care workers such as a decreased adherence with infection control measures as hand hygiene, stress and fatigue of caregivers, an excessive workload, a high nurse turnover or their absenteeism, the work schedules, as well as, by individual factors such as, the work experience, age, and the organizational climate as root causes.

In this research the following factors will be taken into account:

* at the organizational level: the type and size of hospital departments (in number of beds and in number of caregivers), the hourly organization of the staff, the number of caregivers by professional category for each shift in 24h;
* at the hospital department level: nurse absenteeism and turnover rates, safety culture, healthcare-associated infections rates, the rate of blood exposure accidents among caregivers, hand hygiene compliance rates;
* at the level of caregivers: age, sex, personal situation, number of young children, occupation, the position held, work experience, work schedules, stress and fatigue levels, blood exposure accidents, excessive work-related commitment, the social support from coworkers and from supervisors, current state of health, absences due to health reasons including absences due to accidents at work or for work-related illness, etc.

ELIGIBILITY:
Inclusion Criteria:

For hospital departments:

- acute-care departments among medicine (including geriatrics and pediatrics), surgery, gynecology, obstetrics, intensive care, having at least 30 caregivers (medical and paramedical staff) working for the department.

Non-inclusion criteria for hospital departments:

* departments having low care activity such as the long-term care, follow-up care, and rehabilitation, psychiatric departments
* hospitals departments for which a closure or restructuring is in progress or planned within 15 months of the start of the investigation.

Inclusion criteria for caregivers:

- statutory and contractual caregivers (nursing assistants, registered nurses, doctors or midwives) working at least at 0.5 full-time-equivalent who will be present at the time of inclusion visit, and having expressed their non-opposition to participate in the study.

Non-inclusion criteria for caregivers:

* all interim (temporary) caregivers, medical students or interns or residents, as likely to change the hospital department during the investigation;
* caregivers (medical or paramedical) whose departure is planned within 15 months of the start of the survey (e.g. pregnant women, caregivers whose retirement is imminent, caregivers waiting for reassignment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population is the medical (doctors, midwives) and paramedical (nurses' aides, registered nurses, specialized nurses and head nurses) staff, working in hospital departments drawn at random among five volunteer hospital centers in Paris, and who will be present at the time of investigator's passage, at a date drawn at random during the inclusion phase.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Infectious risk in the participating hospital departments | at Day 0
  Incidence rate of blood exposure accidents (BEA) at t0 in the participating hospital departments.
  The BEA rate will be expressed as the report of the number of declared BEAs on the total number of caregivers interviewed during these periods.
Infectious risk in the participating hospital departments | at Months 4
  Incidence rate of blood exposure accidents (BEA) at t1 in the participating hospital departments.
  The BEA rate will be expressed as the report of the number of declared BEAs on the total number of caregivers interviewed during these periods.
Infectious risk in the participating hospital departments | at Months 8
  Incidence rate of blood exposure accidents (BEA) at t2 in the participating hospital departments.
  The BEA rate will be expressed as the report of the number of declared BEAs on the total number of caregivers interviewed during these periods.
Infectious risk in the participating hospital departments | at Months 12
  Incidence rate of blood exposure accidents (BEA) at t3 in the participating hospital departments.
  The BEA rate will be expressed as the report of the number of declared BEAs on the total number of caregivers interviewed during these periods.
Incidence rate of healthcare-associated infections (HAI) | at Day 0
  - The incidence rate of healthcare-associated infections (HAIs) among inpatients in the participating hospitals departments at t0. Data from the Program for Medicalization of Information Systems (PMSI) of each hospital center will be used as data source. The rate will be expressed as the report of the number of HAIs, listed in the PMSI as significant associated diagnosis, on the total number of hospitalized patients.
Incidence rate of healthcare-associated infections (HAI) | at Months 4
  - The incidence rate of healthcare-associated infections (HAIs) among inpatients in the participating hospitals departments at t0
Incidence rate of healthcare-associated infections (HAI) | at Months 8
  - The incidence rate of healthcare-associated infections (HAIs) among inpatients in the participating hospitals departments at t2
Incidence rate of healthcare-associated infections (HAI) | at Months 12
  - The incidence rate of healthcare-associated infections (HAIs) among inpatients in the participating hospitals departments at t3

SECONDARY OUTCOMES:
Stress level of caregivers | at Day 0
  Stress level of caregivers surveyed in the participating hospital departments measured by validated scales (PSS-10 scale). The French version of the 10-item perceived stress scale scoring (PSS-10) will be used to measure the stress at the individual level. Scores ranging from 27 to 40 on the PSS-10 will be considered as high stress levels.
Stress level of caregivers | at Months 4
  Stress level of caregivers surveyed in the participating hospital departments measured by validated scales (PSS-10 scale). The French version of the 10-item perceived stress scale scoring (PSS-10) will be used to measure the stress at the individual level. Scores ranging from 27 to 40 on the PSS-10 will be considered as high stress levels.
Stress level of caregivers | at Months 8
  Stress level of caregivers surveyed in the participating hospital departments measured by validated scales (PSS-10 scale). The French version of the 10-item perceived stress scale scoring (PSS-10) will be used to measure the stress at the individual level. Scores ranging from 27 to 40 on the PSS-10 will be considered as high stress levels.
Stress level of caregivers | at Months 12
  Stress level of caregivers surveyed in the participating hospital departments measured by validated scales (PSS-10 scale). The French version of the 10-item perceived stress scale scoring (PSS-10) will be used to measure the stress at the individual level. Scores ranging from 27 to 40 on the PSS-10 will be considered as high stress levels.
Fatigue level of caregivers | at Day 0
  Fatigue level of caregivers surveyed in the participating hospital departments measured by validated Pichot fatigue questionnaire. The Pichot fatigue questionnaire will be used to measure it at the individual level. Scores ranging from 22 to 32 on the Pichot fatigue questionnaire will be considered as high fatigue levels.
Fatigue level of caregivers | at Months 4
  Fatigue level of caregivers surveyed in the participating hospital departments measured by validated Pichot fatigue questionnaire. The Pichot fatigue questionnaire will be used to measure it at the individual level. Scores ranging from 22 to 32 on the Pichot fatigue questionnaire will be considered as high fatigue levels.
Fatigue level of caregivers | at Months 8
  Fatigue level of caregivers surveyed in the participating hospital departments measured by validated Pichot fatigue questionnaire. The Pichot fatigue questionnaire will be used to measure it at the individual level. Scores ranging from 22 to 32 on the Pichot fatigue questionnaire will be considered as high fatigue levels.
Fatigue level of caregivers | at Months 12
  Fatigue level of caregivers surveyed in the participating hospital departments measured by validated Pichot fatigue questionnaire. The Pichot fatigue questionnaire will be used to measure it at the individual level. Scores ranging from 22 to 32 on the Pichot fatigue questionnaire will be considered as high fatigue levels.
Hand hygiene compliance rate in the participating hospital departments, measured via the GREPHH quick-audit system | at Day 0
  It will be measured as the number of hand hygiene observation divided by the total number of hand hygiene opportunities according to the GREPHH's quick-audit system. The quick-audits will be carried out in each participating hospital department with the cooperation of the hygiene team of each center, on a given day chosen at random.
Hand hygiene compliance rate in the participating hospital departments, measured via the GREPHH quick-audit system | at Months 4
  It will be measured as the number of hand hygiene observation divided by the total number of hand hygiene opportunities according to the GREPHH's quick-audit system. The quick-audits will be carried out in each participating hospital department with the cooperation of the hygiene team of each center, on a given day chosen at random.
Hand hygiene compliance rate in the participating hospital departments, measured via the GREPHH quick-audit system | at Months 8
  It will be measured as the number of hand hygiene observation divided by the total number of hand hygiene opportunities according to the GREPHH's quick-audit system. The quick-audits will be carried out in each participating hospital department with the cooperation of the hygiene team of each center, on a given day chosen at random.
Hand hygiene compliance rate in the participating hospital departments, measured via the GREPHH quick-audit system | at Months 12
  It will be measured as the number of hand hygiene observation divided by the total number of hand hygiene opportunities according to the GREPHH's quick-audit system. The quick-audits will be carried out in each participating hospital department with the cooperation of the hygiene team of each center, on a given day chosen at random.
Caregiver absenteeism rate in the participating hospital departments (absences due to health reasons including absences due to accidents at work or for work-related illness), measured on the basis of human resources data | at Day 0
  The caregiver absenteeism rate in the participating hospital departments (absences due to health reasons including absences due to accidents at work or for work-related illness), measured on the basis of human resources data, at t0, t1 (t0 + 4 month), t2 (t0 + 8 month), t3 ((t0 + 12 month). It will be expressed as the percentage of the overall days (or hours) that a member of staff could have worked, had they not been absent.
Caregiver absenteeism rate in the participating hospital departments (absences due to health reasons including absences due to accidents at work or for work-related illness), measured on the basis of human resources data | at Months 4
  The caregiver absenteeism rate in the participating hospital departments (absences due to health reasons including absences due to accidents at work or for work-related illness), measured on the basis of human resources data, at t0, t1 (t0 + 4 month), t2 (t0 + 8 month), t3 ((t0 + 12 month). It will be expressed as the percentage of the overall days (or hours) that a member of staff could have worked, had they not been absent.
Caregiver absenteeism rate in the participating hospital departments (absences due to health reasons including absences due to accidents at work or for work-related illness), measured on the basis of human resources data | at Months 8
  The caregiver absenteeism rate in the participating hospital departments (absences due to health reasons including absences due to accidents at work or for work-related illness), measured on the basis of human resources data, at t0, t1 (t0 + 4 month), t2 (t0 + 8 month), t3 ((t0 + 12 month). It will be expressed as the percentage of the overall days (or hours) that a member of staff could have worked, had they not been absent.
Caregiver absenteeism rate in the participating hospital departments (absences due to health reasons including absences due to accidents at work or for work-related illness), measured on the basis of human resources data | at Months 12
  The caregiver absenteeism rate in the participating hospital departments (absences due to health reasons including absences due to accidents at work or for work-related illness), measured on the basis of human resources data, at t3.
Caregiver turnover rate in the participating hospitals departments, measured on the basis of human resources data | at Day 0
  The caregiver turnover rate will be expressed as the total number of caregiver departures divided by the total number of caregivers at t0.
Caregiver turnover rate in the participating hospitals departments, measured on the basis of human resources data | at Months 4
  The caregiver turnover rate will be expressed as the total number of caregiver departures divided by the total number of caregivers at t1.
Caregiver turnover rate in the participating hospitals departments, measured on the basis of human resources data | at Months 8
  The caregiver turnover rate will be expressed as the total number of caregiver departures divided by the total number of caregivers at t2.
Caregiver turnover rate in the participating hospitals departments, measured on the basis of human resources data | at Months 12
  The caregiver turnover rate will be expressed as the total number of caregiver departures divided by the total number of caregivers at t3.
Ergonomic analysis of the activity on 2 participating hospital departments per hospital center and with voluntary caregivers, based on a qualitative approach consisting on interviews and observations | at Day 0
  An ergonomic analysis of the activity on 2 participating hospital departments per hospital center and with voluntary caregivers, based on a qualitative approach consisting of interviews and observations of the real work of workers, through the methodology the ergonomics of the activity at t0, The data collected during the interviews will be analyzed by thematic analysis of the content and frequency of appearance of the categories determined from a standardized survey grid and the corpus of verbalizations. The data collected during the observations of the real work will be treated through an activity analysis grid that aims to identify and analyze the operating modes, the regulation strategies and the conflicts of goals and the arbitrations of the caregivers.
Ergonomic analysis of the activity on 2 participating hospital departments per hospital center and with voluntary caregivers, based on a qualitative approach consisting on interviews and observations | at Months 4
  An ergonomic analysis of the activity on 2 participating hospital departments per hospital center and with voluntary caregivers, based on a qualitative approach consisting of interviews and observations of the real work of workers, through the methodology the ergonomics of the activity at t1.
Ergonomic analysis of the activity on 2 participating hospital departments per hospital center and with voluntary caregivers, based on a qualitative approach consisting on interviews and observations | at Months 8
  An ergonomic analysis of the activity on 2 participating hospital departments per hospital center and with voluntary caregivers, based on a qualitative approach consisting of interviews and observations of the real work of workers, through the methodology the ergonomics of the activity at t2.
Ergonomic analysis of the activity on 2 participating hospital departments per hospital center and with voluntary caregivers, based on a qualitative approach consisting on interviews and observations | at Months 12
  An ergonomic analysis of the activity on 2 participating hospital departments per hospital center and with voluntary caregivers, based on a qualitative approach consisting of interviews and observations of the real work of workers, through the methodology the ergonomics of the activity at t3.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal ASTAGNEAU, MD-PhD, Principal Investigator — CPias Ile-de-France (AP-HP)
Locations (1):
- Assistance publique - Hôpitaux de Paris, Paris, France